CLINICAL TRIAL: NCT04625465
Title: Proximal Effects of Alcohol on Same-Sex Intimate Partner Violence
Acronym: PASSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: University at Buffalo (Other); University of Louisville (Other)
Responsible Party: Principal Investigator, Dominic Parrott, Principal Investigator, Georgia State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA025995 (NIH)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Consumption; Violence, Domestic; Stress, Psychological; Aggression
Keywords: sexual minority; gender minority
MeSH Terms: conditions — Alcohol Drinking; Stress, Psychological; Aggression

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled into a measurement burst daily diary design comprised of four 14-day bursts of daily surveys with three 14-day intervals that do not include daily surveys. There are three intervention conditions: (A) no intervention; (B) attention-control text messaging; or (C) CBT text messaging intervention. Between bursts 1 and 2 (Interval 1), all participants will be assigned to condition A (no intervention) such that all will complete the first two bursts (28 days) before receiving an intervention. Between bursts 2 and 3 (Interval 2) and bursts 3 and 4 (Interval 3), couples will be randomized to one of the following eight patterns of conditions: AA, AB, AC, BA, BB, BC, CA, or CB. There is no "CC" condition because the CBT intervention is not intended to be given in multiple two-week intervals.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- No Intervention, No Intervention (AA) (No Intervention): Participants do not receive text messages during Interval 2 or Interval 3.
- No Intervention, Attention-Control Texts (AB) (Active Comparator): Participants do not receive text messages during Interval 2. Participants receive attention control text messages during Interval 3.
  Interventions: Behavioral: Attention Control Text Messaging
- No Intervention, CBT Texts (AC) (Experimental): Participants do not receive text messages during Interval 2. Participants receive CBT text messages during Interval 3.
  Interventions: Behavioral: CBT Text Messaging
- Attention-Control Texts, No Intervention (BA) (Active Comparator): Participants receive attention control text messages during Interval 2. Participants do not receive text messages during Interval 3.
  Interventions: Behavioral: Attention Control Text Messaging
- Attention-Control Texts, Attention-Control Texts (BB) (Active Comparator): Participants receive attention control text messages during Interval 2. Participants receive attention control text messages during Interval 3.
  Interventions: Behavioral: Attention Control Text Messaging
- Attention-Control Texts, CBT Texts (BC) (Experimental): Participants receive attention control text messages during Interval 2. Participants receive CBT text messages during Interval 3.
  Interventions: Behavioral: CBT Text Messaging; Behavioral: Attention Control Text Messaging
- CBT Texts, No Intervention (CA) (Experimental): Participants receive CBT text messages during Interval 2. Participants do not receive text messages during Interval 3.
  Interventions: Behavioral: CBT Text Messaging
- CBT Texts, Attention-Control Texts (CB) (Experimental): Participants receive CBT text messages during Interval 2. Participants receive attention control text messages during Interval 3.
  Interventions: Behavioral: CBT Text Messaging; Behavioral: Attention Control Text Messaging

INTERVENTIONS:
Behavioral: CBT Text Messaging — Over a 14 day period, participants will receive two text messages per day (one at 8 a.m. and one at 4 p.m.). They will receive hourly reminders for four hours or until the message is read. Participants receive the same messages in the same order, with content equally distributed across the four content areas (i.e., psychoeducation regarding effects of stress, distress tolerance, emotion regulation, alcohol reduction).
  Arms: Attention-Control Texts, CBT Texts (BC); CBT Texts, Attention-Control Texts (CB); CBT Texts, No Intervention (CA); No Intervention, CBT Texts (AC)
Behavioral: Attention Control Text Messaging — Over a 14 day period, participants will receive two text messages per day (one at 8 a.m. and one at 4 p.m.). They will receive hourly reminders for four hours or until the message is read. Participants receive the same messages in the same order. All texts will be supportive messages which express empathy and unconditional positive regard and provide support for dealing with stressors. These messages will be nondirective and will not include any CBT skill suggestions.
  Arms: Attention-Control Texts, Attention-Control Texts (BB); Attention-Control Texts, CBT Texts (BC); Attention-Control Texts, No Intervention (BA); CBT Texts, Attention-Control Texts (CB); No Intervention, Attention-Control Texts (AB)

SUMMARY:
We will recruit sexual and gender minority couples to complete 56 days of daily surveys in order to evaluate (1) the impact of COVID-19 stress and sexual and gender minority stress on heavy episodic drinking and intimate partner violence (IPV) perpetration, and (2) a brief, mobile-phone delivered text messaging intervention to mitigate the effects of these stressors. This project has high potential to inform how pandemic stress contributes to etiological models of alcohol-related IPV perpetration in sexual and gender minority couples and inform a culturally-sensitive, low burden, and easy to disseminate intervention to mitigate these effects critical during a pandemic when access to care is limited.

ELIGIBILITY:
Inclusion Criteria (applies to both partners):

* Both partners must identify as cisgender and sexual minority or at least one partner must identify as a gender minority (i.e., one's gender identity is non-congruent with their sex assigned at birth)
* 21 years or older
* In an intimate relationship lasting at least one month in which there are at least 2 days of face-to-face contact each week
* Consumption of 4 (assigned female at birth) or 5 (assigned male at birth) alcoholic drinks on at least three days in the past year

Exclusion Criteria:

* Seeking treatment or being in recovery for an alcohol or substance use disorder.
* Endorsement of severe physical IPV (e.g., use of a weapon) in the past year.
* Women who self-report that they are trying to get pregnant, that they are currently pregnant, or that they are currently breastfeeding .

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic J Parrott, Ph.D., Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
After the grant period, access to the data will be provided through the Inter-University Consortium for Political and Social Research (ICPSR). Users will be required to agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data source and funders. One year after the study is completed, all data will be compiled and organized into a single repository at ICPSR. Data will be made publicly available through ICPSR's website.
Time Frame: One year after the study is completed, all data will be compiled and organized into a single repository at ICPSR.
Access Criteria: Users will be required to agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data source and funders.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Started | 40 | 38 | 76 | 40 | 40 | 80 | 80 | 80
Completed | 36 | 36 | 71 | 36 | 36 | 78 | 80 | 80
Not Completed | 4 | 2 | 5 | 4 | 4 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 4 | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant (n=1) dropped from the analysis because the other dyad member was lost to follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB) | Total
Number analyzed (Participants) | 36 | 36 | 70 | 36 | 36 | 78 | 80 | 80 | 452
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participant's self-reported chronological age measured in years
  Years | 32.69 (10.92) | 27.28 (4.41) | 29.81 (7.92) | 27.47 (5.07) | 28.61 (9.77) | 28.86 (7.04) | 30.36 (8.66) | 28.25 (6.87) | 29.21 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants] — Prompt: What sex were you assigned at birth?
  Participants
    Female | 29 | 25 | 54 | 25 | 23 | 60 | 52 | 59 | 327
    Male | 7 | 11 | 16 | 11 | 13 | 18 | 28 | 21 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants] — Prompt: How do you describe your race (Select all that apply)?
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
    Asian | 6 | 2 | 2 | 2 | 2 | 4 | 1 | 4 | 23
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Black or African American | 11 | 5 | 5 | 3 | 6 | 17 | 16 | 12 | 75
    White | 19 | 27 | 62 | 26 | 24 | 51 | 59 | 61 | 329
    More than one race | 0 | 1 | 0 | 2 | 4 | 4 | 4 | 3 | 18
    Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Prompt: How do you describe your ethnicity?
  Participants
    Hispanic or Latino | 4 | 5 | 9 | 4 | 3 | 10 | 9 | 9 | 53
    Not Hispanic or Latino | 32 | 31 | 61 | 32 | 33 | 68 | 71 | 71 | 399
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gender minority status [Count of Participants; unit: Participants] — Indicator of correspondence between self-reported sex assigned at birth and answer to the following prompt: How do you describe your gender (select all that apply)?
  Participants
    Gender minority | 10 | 13 | 25 | 11 | 13 | 25 | 24 | 24 | 145
    Cisgender | 26 | 23 | 45 | 25 | 23 | 53 | 56 | 56 | 307

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use (Burst 1)
Description: Proportion of reporting days on which alcohol was consumed
Time Frame: Burst 1, Daily for 14 days
Population: 452 participants, across all arms, had reported outcome for Burst 1. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 36 | 70 | 36 | 36 | 78 | 80 | 80
Proportion of reporting days | .45 (.29) | .40 (.23) | .41 (.30) | .31 (.27) | .45 (.27) | .41 (.23) | .44 (.31) | .42 (.28)

2. Primary Outcome: Alcohol Use (Burst 2)
Description: Proportion of reporting days on which alcohol was consumed
Time Frame: Burst 2, Daily for 14 days
Population: Only 448 of 452 participants, across all arms, had reported outcome for Burst 2. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 33 | 70 | 36 | 36 | 77 | 80 | 80
Proportion of reporting days | .49 (.31) | .42 (.21) | .41 (.29) | .30 (.26) | .42 (.27) | .38 (.24) | .48 (.32) | .42 (.29)

3. Primary Outcome: Alcohol Use (Burst 3)
Description: Proportion of reporting days on which alcohol was consumed
Time Frame: Burst 3, Daily for 14 days
Population: Only 429 of 452 participants, across all arms, had reported outcome for Burst 3. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 35 | 33 | 63 | 35 | 35 | 78 | 77 | 73
Proportion of reporting days | .45 (.31) | .41 (.24) | .42 (.30) | .35 (.27) | .39 (.27) | .39 (.29) | .43 (.32) | .36 (.28)

4. Primary Outcome: Alcohol Use (Burst 4)
Description: Proportion of reporting days on which alcohol was consumed
Time Frame: Burst 4, Daily for 14 days
Population: Only 435 of 452 participants, across all arms, had reported outcome for Burst 4. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 35 | 32 | 66 | 35 | 35 | 76 | 79 | 77
Proportion of reporting days | .45 (.35) | .43 (.26) | .41 (.32) | .34 (.27) | .40 (.29) | .34 (.24) | .41 (.36) | .36 (.29)

5. Primary Outcome: Intimate Partner Violence (IPV) Perpetration (Burst 1)
Description: Proportion of reporting days on which IPV perpetration occurred
Time Frame: Burst 1, Daily for 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 36 | 70 | 36 | 36 | 78 | 80 | 80
Proportion of reporting days | .019 (.034) | .035 (.066) | .031 (.058) | .031 (.062) | .017 (.036) | .024 (.050) | .022 (.051) | .041 (.070)

6. Primary Outcome: IPV Perpetration (Burst 2)
Description: Proportion of reporting days on which IPV perpetration occurred
Time Frame: Burst 2, Daily for 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 33 | 70 | 36 | 36 | 77 | 80 | 80
Proportion of reporting days | .047 (.113) | .013 (.039) | .015 (.041) | .026 (.057) | .018 (.038) | .026 (.046) | .025 (.050) | .035 (.066)

7. Primary Outcome: IPV Perpetration (Burst 3)
Description: Proportion of reporting days on which IPV perpetration occurred
Time Frame: Burst 3, Daily for 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 35 | 33 | 63 | 35 | 35 | 78 | 77 | 73
Proportion of reporting days | .042 (.101) | .049 (.081) | .018 (.043) | .019 (.056) | .015 (.050) | .021 (.050) | .014 (.041) | .053 (.139)

8. Primary Outcome: IPV Perpetration (Burst 4)
Description: Proportion of reporting days on which IPV perpetration occurred
Time Frame: Burst 4, Daily for 14 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Proportion of reporting days
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 35 | 32 | 66 | 35 | 35 | 76 | 79 | 77
Proportion of reporting days | .042 (.135) | .020 (.039) | .017 (.048) | .014 (.032) | .045 (.139) | .026 (.069) | .011 (.036) | .033 (.070)

9. Secondary Outcome: Sexual Minority Stress (Burst 1)
Description: Total daily count across 15 daily sexual minority stress (SMS) indicators
Time Frame: Burst 1, Daily for 14 days
Population: Only 451 of 452 participants, across all arms, had reported outcome for Burst 1. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of SMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 36 | 70 | 36 | 36 | 78 | 79 | 80
Average daily count of SMS indicators | .48 (.53) | .54 (.56) | .55 (.71) | .59 (.64) | .32 (.37) | .42 (.57) | .50 (1.23) | .58 (.82)

10. Secondary Outcome: Sexual Minority Stress (Burst 2)
Description: Total daily count across 15 daily sexual minority stress (SMS) indicators
Time Frame: Burst 2, Daily for 14 days
Population: Only 447 of 452 participants, across all arms, had reported outcome for Burst 2. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of SMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 33 | 70 | 36 | 36 | 77 | 79 | 80
Average daily count of SMS indicators | .39 (.46) | .32 (.40) | .53 (.62) | .42 (.65) | .32 (.36) | .36 (.69) | .43 (1.26) | .37 (.49)

11. Secondary Outcome: Sexual Minority Stress (Burst 3)
Description: Total daily count across 15 daily sexual minority stress (SMS) indicators
Time Frame: Burst 3, Daily for 14 days
Population: Only 428 of 452 participants, across all arms, had reported outcome for Burst 3. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of SMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 35 | 33 | 63 | 35 | 35 | 78 | 76 | 73
Average daily count of SMS indicators | .31 (.39) | .29 (.35) | .41 (.69) | .42 (.65) | .31 (.44) | .30 (.59) | .31 (1.02) | .30 (.53)

12. Secondary Outcome: Sexual Minority Stress (Burst 4)
Description: Total daily count across 15 daily sexual minority stress (SMS) indicators
Time Frame: Burst 4, Daily for 14 days
Population: Only 434 of 452 participants, across all arms, had reported outcome for Burst 4. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of SMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 35 | 32 | 66 | 35 | 35 | 76 | 78 | 77
Average daily count of SMS indicators | .34 (.63) | .37 (.44) | .34 (.48) | .32 (.53) | .39 (.72) | .33 (.74) | .26 (1.16) | .30 (.38)

13. Secondary Outcome: Gender Minority Stress (Burst 1)
Description: Total daily count across 14 daily gender minority stress (GMS) indicators
Time Frame: Burst 1, Daily for 14 days
Population: Only 162 of 452 participants, across all arms, had reported outcome for Burst 1. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of GMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 10 | 14 | 28 | 12 | 14 | 28 | 27 | 29
Average daily count of GMS indicators | .80 (.79) | .73 (.50) | 1.17 (1.04) | 1.13 (.88) | .73 (.44) | 1.09 (.87) | .94 (2.17) | 1.14 (.99)

14. Secondary Outcome: Gender Minority Stress (Burst 2)
Description: Total daily count across 14 daily gender minority stress (GMS) indicators
Time Frame: Burst 2, Daily for 14 days
Population: Only 162 of 452 participants, across all arms, had reported outcome for Burst 2. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of GMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 10 | 14 | 28 | 12 | 14 | 28 | 28 | 28
Average daily count of GMS indicators | .82 (1.04) | .64 (.48) | 1.05 (1.09) | .73 (1.07) | .91 (.74) | .95 (.85) | .97 (2.14) | .95 (.92)

15. Secondary Outcome: Gender Minority Stress (Burst 3)
Description: Total daily count across 14 daily gender minority stress (GMS) indicators
Time Frame: Burst 3, Daily for 14 days
Population: Only 145 of 452 participants, across all arms, had reported outcome for Burst 3. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of GMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 10 | 14 | 21 | 11 | 13 | 28 | 25 | 23
Average daily count of GMS indicators | .50 (.77) | .80 (.82) | .77 (1.02) | .73 (1.16) | .73 (.63) | .98 (1.06) | .89 (2.13) | .87 (.98)

16. Secondary Outcome: Gender Minority Stress (Burst 4)
Description: Total daily count across 14 daily gender minority stress (GMS) indicators
Time Frame: Burst 4, Daily for 14 days
Population: Only 153 of 452 participants, across all arms, had reported outcome for Burst 4. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of GMS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 10 | 13 | 25 | 11 | 13 | 27 | 26 | 28
Average daily count of GMS indicators | .24 (.42) | .46 (.59) | .70 (.70) | .41 (.53) | .76 (.81) | .93 (1.52) | .88 (2.33) | .65 (.73)

17. Secondary Outcome: COVID Stress (Burst 1)
Description: Average daily count of COVID stress (CS) indicators
Time Frame: Burst 1, Daily for 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average daily count of CS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 36 | 70 | 36 | 36 | 78 | 80 | 80
Average daily count of CS indicators | 1.88 (1.11) | 2.07 (1.07) | 1.81 (.83) | 1.87 (1.00) | 1.61 (.99) | 1.69 (.85) | 1.72 (.98) | 1.84 (1.01)

18. Secondary Outcome: COVID Stress (Burst 2)
Description: Average daily count of COVID stress (CS) indicators
Time Frame: Burst 2, Daily for 14 days
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Average daily count of CS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 36 | 33 | 70 | 36 | 36 | 77 | 79 | 80
Average daily count of CS indicators | 1.88 (1.11) | 2.07 (1.07) | 1.81 (.83) | 1.88 (1.00) | 1.61 (.99) | 1.69 (.85) | 1.72 (.98) | 1.84 (1.01)

19. Secondary Outcome: COVID Stress (Burst 3)
Description: Average daily count of COVID stress (CS) indicators
Time Frame: Burst 3, Daily for 14 days
Population: Only 427 of 452 participants, across all arms, had reported outcome for Burst 3. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of CS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 34 | 33 | 63 | 35 | 35 | 78 | 76 | 73
Average daily count of CS indicators | 2.20 (1.22) | 1.93 (.99) | 1.80 (.79) | 1.88 (1.06) | 1.64 (.97) | 1.70 (.88) | 1.77 (1.01) | 1.85 (1.03)

20. Secondary Outcome: COVID Stress (Burst 4)
Description: Average daily count of COVID stress (CS) indicators
Time Frame: Burst 4, Daily for 14 days
Population: Only 432 of 452 participants, across all arms, had reported outcome for Burst 4. Results data were pre-specified according to the Study Protocol and Statistical Analysis Plan to be assessed in the per-sequence Arms/Groups (e.g., "No Intervention, No Intervention (AA)", "Attention-Control Texts, Attention-Control Texts (BB)", "CBT Texts, Attention-Control Texts (CB)"). Thus, no arms are combined and all results are reported for each arm separately.
Measure: Mean (Standard Deviation); unit: Average daily count of CS indicators
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
Number analyzed (Participants) | 33 | 32 | 66 | 35 | 35 | 76 | 78 | 77
Average daily count of CS indicators | 2.09 (1.25) | 2.00 (1.03) | 1.87 (.91) | 1.82 (1.03) | 1.65 (.97) | 1.65 (.80) | 1.71 (.99) | 1.87 (1.02)

21. Primary Outcome: Alcohol Use --> IPV Perpetration (Pre-Intervention)
Description: Odds ratio (OR) of IPV perpetration corresponding to alcohol use (versus non-use).
  Estimated using a multilevel logistic regression of daily IPV perpetration on alcohol use (Level 1) nested within participant (Level 2).
Time Frame: Bursts 1 and 2 (daily for 14 x 2 days)
Population: The Study Aims, as funded, sought to compare combinations of intervention arms. Thus, per this proposed analytic strategy, arms corresponding to control or intervention status were combined as appropriate to permit the analysis of hypothesized intervention main effects.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- No Intervention and Attention Control (AA, AB, BA, BB): See Protocol for description of intervention conditions AA, AB, BA, and BB.
- CBT Texts Intervention (AC, BC, CA, CB): See Protocol for description of intervention conditions AC, BC, CA, and CB.
Arm/Group | No Intervention and Attention Control (AA, AB, BA, BB) | CBT Texts Intervention (AC, BC, CA, CB)
Number analyzed (Participants) | 144 | 308
Odds Ratio | 1.26 [.87 to 1.82] | 1.32 [.95 to 1.82]
Statistical Analysis 1: Comparison: No Intervention and Attention Control (AA, AB, BA, BB) vs CBT Texts Intervention (AC, BC, CA, CB); Multilevel logistic regression of daily IPV perpetration on alcohol use (Level 1) nested within participant (Level 2) with interaction between alcohol use and CBT Intervention. Testing the difference in odds ratio between groups 1 (No Intervention and Attention Control ) and 2 (CBT Texts Intervention) H0: OR1 = OR2; Test type: Other; p = .869, Multilevel logistic regression; Difference in the log odds ratios = .042

22. Primary Outcome: Alcohol Use --> IPV Perpetration (Post-Intervention)
Description: as for outcome 21
Time Frame: Bursts 3 and 4 (daily for 14 x 2 days)
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | No Intervention and Attention Control (AA, AB, BA, BB) | CBT Texts Intervention (AC, BC, CA, CB)
Number analyzed (Participants) | 144 | 308
Odds Ratio | 1.48 [.91 to 2.41] | 1.06 [.82 to 1.37]
Statistical Analysis 1: Comparison: No Intervention and Attention Control (AA, AB, BA, BB) vs CBT Texts Intervention (AC, BC, CA, CB); [analysis description as in outcome 21, analysis 1]; Test type: Other; p = .210, Multilevel logistic regression; Difference in the log odds ratios = -.32

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time after participants completed the baseline survey until they time they completed the fourth burst of daily diaries (i.e., approximately 14 weeks).
Description: This project's definition of an adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definition.
Arm/Group | No Intervention, No Intervention (AA) | No Intervention, Attention-Control Texts (AB) | No Intervention, CBT Texts (AC) | Attention-Control Texts, No Intervention (BA) | Attention-Control Texts, Attention-Control Texts (BB) | Attention-Control Texts, CBT Texts (BC) | CBT Texts, No Intervention (CA) | CBT Texts, Attention-Control Texts (CB)
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/38 | 0/76 | 0/40 | 0/40 | 0/80 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/38 | 0/76 | 0/40 | 0/40 | 0/80 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/76 | 0/40 | 0/40 | 0/80 | 0/80 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention, No Intervention (AA) (N=40) | No Intervention, Attention-Control Texts (AB) (N=38) | No Intervention, CBT Texts (AC) (N=76) | Attention-Control Texts, No Intervention (BA) (N=40) | Attention-Control Texts, Attention-Control Texts (BB) (N=40) | Attention-Control Texts, CBT Texts (BC) (N=80) | CBT Texts, No Intervention (CA) (N=80) | CBT Texts, Attention-Control Texts (CB) (N=80)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The participant's death was not related to the intervention. The participant's partner reported the participant's death; however, we were not informed of the cause of death. Thus, we selected "General Disorders" as the organ system affected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04625465/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT04625465/ICF_002.pdf